CLINICAL TRIAL: NCT01384461
Title: An Open-label, Multicenter Non-interventional Trial to Evaluate Safety, Tolerability and Efficacy of Tocilizumab in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: An Observational Study of RoActemra/Actemra (Tocilizumab) in Combination With Methotrexate in Patients With Rheumatoid Arthritis (ACTIVATE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25503
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the safety, tolerability and efficacy of RoActemra/Actemra (tocilizumab) in combination with methotrexate in patients with moderate to severe rheumatoid arthritis. Data will be collected for 12 months from patients initiated on treatment with RoActemra/Actemra (8 mg/kg intravenously every 4 weeks) and methotrexate (weekly dose at the discretion of the physician).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe rheumatoid arthritis
* RoActemra/Actemra treatment initiated by rheumatologist in an Arthritis Center for (up to 2 months prior to study entry)

Exclusion Criteria:

* History of severe allergic or anaphylactic reactions or known hypersensitivity to any component of the drug
* Active, severe infection or history of recurrent clinically significant infection
* Pregnancy
* Treatment with an investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before baseline visit
* Methotrexate intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe rheumatoid arthritis initiated on treatment with RoActemra/Actemra in combination with methotrexate
Sampling Method: Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 12 months

SECONDARY OUTCOMES:
Efficacy: Disease Activity Score (DAS 28) | 12 months
Pain: Visual Analogue Scale (VAS) pain scale | 12 months
Physical Function: Health Assessments Questionnaire (HAQ) | 12 months
Incidence of patients with all-cause discontinuation of tocilizumab | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (17):
- Hungary (17):
  - Budapest
  - Debrecen
  - Eger
  - Esztergom
  - Győr
  - Gyula
  - Hévíz
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Veszprém